CLINICAL TRIAL: NCT03040349
Title: Evaluation of the Primary Care Tobacco Treatment TrAining Network in Greece & Cyprus
Brief Title: Tobacco Treatment TrAining Network in Greece & Cyprus
Acronym: TiTAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Crete (Other)
Collaborators: Ottawa Heart Institute Research Corporation (Other); Aristotle University Of Thessaloniki (Other); Global Bridges Healthcare Alliance for Tobacco Dependence Treatment (Mayo Clinic) (Unknown); University of Ioannina (Other); University of Nicosia (Other); Pfizer Grants for Learning and Change (Unknown)
Responsible Party: Principal Investigator, Christor Lionis, Professor, Clinic of Social and Family Medicine, Dept Medicine, University of Crete
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELKE4599
Record Dates: First submitted 2017-01-30; First posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Tobacco Use
Keywords: primary care; greece; cyprus; tobacco use treatment; evidence-based guidelines
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TiTAN Intervention (Experimental): The TiTAN Crete program has adapted the existing curricula and resources originally developed at the University of Ottawa Heart Institute and which are specific to primary practice settings. To facilitate maximum uptake the intervention program was adapted to reflect: language; cultural appropriateness; local patient beliefs and attitudes regarding tobacco-use and cessation; local social and clinical norms; provider perceptions surrounding 5As delivery; and, practice characteristics. The TiTAN multi-component training includes: 1) a 1-day foundational tobacco treatment training program for general practitioners, 2) the dissemination of provider and patient tools, and 3) E-blasts and webinars to supplement skills development and continuing medical education through e-learning.
  Interventions: Behavioral: Training; Behavioral: Provider and Patient Tools; Behavioral: E-blast and Webinars

INTERVENTIONS:
Behavioral: Training — The training program consists of a one-day core session addressing tobacco use with patients in the context of a busy primary care practice setting.The curriculum design was designed to be 2/3 theory and 1/3 practical. The program employs teaching techniques including role-play and case-study approaches known to enhance practice change.
Behavioral: Provider and Patient Tools — Provider and patient tools were translated and adapted for use in primary care settings in Greece. A tool kit of resources will be distributed to providers which includes: patient tobacco use survey; provider consult form; provider medication reference sheet; patient quit plan booklet; and, waiting room posters. The provider consult form uses a checklist style set-up and provides real-time reminders for conducting an initial smoking cessation visit and follow-up appointments. The TiTAN Crete tools are available online at www.titan.uoc.gr
Behavioral: E-blast and Webinars — In order to develop the network and continue to provide training opportunities for skills development we will develop a communication platform via an email list-serv to proactively communicate with providers who participate in the TiTAN program. A quarterly e-blast will be sent to all health care professionals involved in the TiTAN program. The e-blast will address the latest evidence-base practice, and skill development. Links to videos will also be provided. A webinar series will be scheduled to cover topics identified as interest by the primary health care providers. The webinar series will also be linked the Global Bridges EPACTT project.

SUMMARY:
The overall aim of the TiTAN Greece & Cyprus project is to expand the Global Bridges Tobacco Treatment Training Network in the WHO Europe region through a focus on primary health care providers in Greece and Cyprus. A robust evaluation will be conducted alongside the TiTAN program. A pre-post evaluation will be used to examine the impact on the TiTAN program on:

1. Provider engagement (number of providers attending training), number of local champions;
2. Provider knowledge, beliefs, perceived behavioral control, and intentions related to the delivery of tobacco treatment;
3. Rates of evidence-based tobacco treatments (5As) are delivered to patients who smoke;
4. Provider satisfaction with training program, resources, and network outreach activity and areas for improvement; and
5. Estimates on the impact on patient-level outcomes including number of patient quit smoking at 1 and 3-month follow-up.

All PHC providers will be surveyed before and after the intervention program is delivered. We will randomly select a sub-sample of providers and will survey patients from their practice before and after the intervention program in order to validate changes in 5As delivery. Qualitative interviews will be completed with a sub-sample of providers at the end of year 1.

DETAILED DESCRIPTION:
Design The evaluation design schema is presented in Appendix B. A pre-post evaluation design will be used. All PHC providers will be surveyed before, immediately following the training session and 3-months after the intervention program is delivered. Additionally, a random sample of providers will be identified from which a cross-sectional sample of eligible smokers from their practice will be surveyed pre- and post-intervention to assess provider performance in the delivery of 5As tobacco treatment intervention. Qualitative interviews will be completed with a sub-sample of providers at the end of year 1.

Procedures

Provider Recruitment An invitation letter will be sent to all GPs and other PHC providers in the target region. We will include both GPs working in private and public practices in the target region. A follow-up phone call will be placed to all providers by a member of the investigative team, one week after the invitation was sent to confirm interest in participation. We will aim to reach all providers with a minimum of three attempts being made to reach all providers before classifying them as "unable to contact". Participating providers will sign an information sheet and consent form.

Provider Pre- and Post-Assessment Survey All participating providers will a complete a survey prior to the foundational training (Time 1) which will assess demographic variables and outcomes of interest. Immediately following the training (Time 2) and 3-months following the training (Time 3), providers will complete follow-up surveys which will re-assess outcomes of interest and satisfaction with the intervention program.

Semi-structured interviews will be conducted with 10 PHC providers at the end of year 1 in order to inform year 2 activities. Providers will be asked to self-identify and will be drawn from all sub-regions. These interviews will be conducted by a trained team member and will be recorded. Key themes will be identified and extracted.

Additionally in order to gain an overall picture of the number of initial and consultations for smoking cessation made by participating providers, we will collect information on basic activities for a 1-year period following the introduction of the training program. A contact log has been created which can be used prospectively by providers and or used retrospectively (ie. chart audit).

Patient-Level Sampling In order to gather information about rates of 5As delivery, a sub-sample of 20 GPs will be randomly selected for patient level data collection. From the sub-sample of randomly selected providers, 16 eligible patients will be recruited before (time 1) and after (time 2) intervention delivery.

Patient-level data collection will be limited to GPs as other health care professionals are likely working alongside the GPs as opposed to a separate practice. Provider eligibility for the patient-level evaluation will include:

1. is a GP working in a public or private primary care practice setting;
2. participation in TiTAN training program;
3. GP has not participated in other smoking cessation training in the previous 2-3 years;
4. sees a minimum of 15 patients per day seen in the practice in order to ensure efficient use of data collection resources; and,
5. located within a reasonable distance from where the training will take place in order to minimize costs associated with travel.

Randomization and Informed Consent Randomization will be stratified by region involved in the present study (Crete, Athens, Ioannina, Thessaloniki, Cyprus) and type of practice (private/public) and years of experience. An independent third party researcher will randomly select GPs from the recruitment list provided for inclusion in the present study. GPs selected for participation in the patient-level sampling will be informed via telephone and asked to sign an informed consent for this component of the study.

Patient Pre-Post Data Collection The pre-intervention assessment will be conducted prior to implementing the intervention program to establish baseline activities of the practice. During the screening period, a research assistant will be located in the clinic waiting room. The research assistant will screen consecutive patients scheduled for an annual exam or non-urgent appointment for eligibility using the study screening form.

Recruitment statistics will be recorded using the recruitment tracking sheet]in order to calculate prevalence of tobacco use (total number of tobacco users/total number of patients), reasons for ineligibility and reasons for non-participation.

Eligible patients who agree to participate in the study will review and sign the study information sheet and consent form and contact sheet with the Research Assistant. Participants will be tracked using the study master list and will be assigned a study ID. Only the study ID will be included on the study survey. Consenting patients will then be given the exit survey to complete at the end of the their visit with their primary care provider. The survey will collect information about whether their physician or another clinician asked about their smoking status (ask); advised them to quit smoking (advise); and provided cessation assistance (assist). The exit survey will also gather socio-demographic and smoking history, beliefs, and intentions.

The post-intervention assessment will involve the collection of data from a second cross-sectional sample of 16 patients approximately 3-months following the implementation of the intervention within the practice. The methods described in the pre-intervention assessment will be repeated at the post-assessment.

ELIGIBILITY:
Inclusion Criteria:

* • are a current smoker (>5 cigarette per day on most days of the week);

  * are 18 years of age or older;
  * are scheduled for an annual exam or non-urgent medical appointment at the primary care clinic;
  * are able to read and/or understand Greek; and,
  * have the mental capacity to provide informed consent and complete study protocols.

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-02 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Provider Performance in the Delivery of Cessation Treatments assessed via patient exit survey | Change between pre-intervention and post intervention (3-months)
  Performance in the delivery of each of the 5As will be assessed via exit interview with eligible patients. The survey will ask participants to respond either "yes" or "no" or "don't know" regarding whether their PHC provider asked them about their smoking status (ask); advised them to quit smoking (advise); assessed their readiness to quit (assess); provided assistance with quitting (assist); prescribed pharmacotherapy, provided self-help materials, and arranged follow-up support

SECONDARY OUTCOMES:
Provider Self-efficacy assessed by questionnaire | Change between pre-intervention and post-training (1-month)
  Provider self-efficacy will be assessed before and after the intervention
Provider knowledge assessed by questionnaire | Change between pre-intervention and post intervention (3-months)
  Provider knowledge of evidence-based tobacco treatment guidelines will be assessed using a brief 15-item knowledge assessment to examine key concepts addressed as part of training. The knowledge assessment has been tested as part of the TiTAN Crte project.

CONTACTS AND LOCATIONS:
Overall Officials: Christos Lionis, MD, PhD, Principal Investigator — University of Crete
Locations (1):
- University of Crete, Heraklion, Crete, Greece

IPD SHARING:
Plan to Share IPD: No